CLINICAL TRIAL: NCT05656300
Title: Unravelling the Invisible Infiltrating Component of Glioblastoma Using MRI and a Strong Iron-like Bloodpool Contrast Medium?
Brief Title: Glioblastoma Imaging Using a Strong Iron-like Bloodpool Contrast Medium?
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Radboud University Medical Center (Other)
Collaborators: ZonMw: The Netherlands Organisation for Health Research and Development (Other)
Responsible Party: Sponsor
Other Study IDs: 83297
Record Dates: First submitted 2022-11-25; First posted 2022-12-19 (Actual); Last update posted 2022-12-19 (Actual); Status verified 2022-11

CONDITIONS: Glioblastoma
MeSH Terms: conditions — Glioblastoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 18 Months
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: MRI scan using USPIO particles — Diagnostic imaging

SUMMARY:
Rationale: Visualization of tumor spread is of crucial importance when treating patients suffering from glioblastoma (GBM) as the success of tumor resection depends strongly on the extent of tumor infiltration. Current MRI protocols, however, cannot visualize the extent the tumor infiltration. The use of non-toxic, non-dangerous ultrasmall superparamagnetic biodegradable iron oxide (USPIO) particles as a very strong blood pool contrast agent could help visualizing this invisible infiltration Objective: To what extent, do GBMs infiltrate healthy brain tissue and can we use ultrasmall superparamagnetic iron oxide particles to visualize co-opting infiltrating tumor cells in an attempt to predict regions of tumor recurrence? Study design: This study concerns a single arm prospective observational study. Study population: Patients diagnosed with suspected glioblastoma. Intervention (if applicable): USPIO neuroimaging Main study parameters/endpoints: The main parameter of this study concerns the feasibility of using of USPIO particles in healthy controls (n=6) and glioblastoma patients (n=15).

Nature and extent of the burden and risks associated with participation, benefit and group relatedness: During this study patients will be intravenously injected with low doses of USPIOs. Risks involved with this procedure include: bruising of the skin after venapunction and allergic reaction to USPIO particles.

The application of USPIO neuroimaging can improve diagnosis of patients with suspected glioblastoma, provide more information on the pathophysiology of growth of glioblastoma lesiosn, the role of neuro-inflammation in these lesions and maybe predict regions of tumor recurrence after treatment.

ELIGIBILITY:
Inclusion Criteria:

* Aged between 18 and 75 years
* Diagnosed with suspected glioblastoma
* Eligible for neurosurgical resection and/or chemoradiation therapy.

Exclusion Criteria:

* Younger than 18 years old
* Patients unfit for surgery or lesions unsuitable for neurosurgical treatment

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Clinicians will recruit men and women diagnosed with a suspected glioblastoma who are scheduled to undergo neurosurgical resection and/or chemoradiation therapy as treatment.
Sampling Method: Non-Probability Sample
Enrollment: 15 (Estimated)
Dates: Start 2023-04-01 (Estimated); Primary Completion 2024-04-01 (Estimated); Study Completion 2025-04-01 (Estimated)

PRIMARY OUTCOMES:
Feasibility study of USPIO neuro-imaging in healthy participants (n=6) | 18 months
  To investigate the dosage of USPIO administration for adequate neuro-imaging (e.g. signal to noise ratio optimization), 6 healthy participants will be included. Obtained images will be reviewed by a panel of radiologists to asses quality and diagnostic performance.

SECONDARY OUTCOMES:
Perform MR imaging of glioblastoma by use of a new Off Road multi-sequence protocol (i.e., T1w, T2w, FLAIR, DWI/DTI, SWI, T1w- and T2*w post-USPIO images) in 15 GBM patients. | 18 months
  To investigate images of glioblastoma lesions after USPIO administration, 15 patients will be included. All imaging will be performed using clinical protocols on a clinical MRI scanning system. Images will be pseudonymized and stored at a safe digital location. Obtained images will be reviewed by a panel of radiologists to asses quality and diagnostic performance.
Analyze the obtained images and characterize brain tissue using both a quantitative and qualitative methodology to delineate regions of tumor infiltration. | 18 months
  Qualitative interpretation of MRI images and quantitative volume of interest (VOI) analysis and vascular density analysis will be used to investigate regions of tumor infiltration. Results will contain sensitivity, specificity, negative predictive value and positive predictive value of the Off-Road multi-sequence protocol in detection of GBM infiltration and prediction of regions of tumor recurrence.

IPD SHARING:
Plan to Share IPD: No